CLINICAL TRIAL: NCT00364117
Title: Remote Presence Timely Discharge Management
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No patients were enrolled
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06.01.052; Intouch Technologies Inc; Horizon Blue Cross Blue Shield
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Patient Discharge
Keywords: 150 discharges; adults; Internal Medicine

INTERVENTIONS:
Behavioral: Timely Discharge (Remote Presence Technology)

SUMMARY:
The purpose of this study is to integrate Remote Presence technology in order to increase the number of timely patient discharges before 11 am from the medical center.

DETAILED DESCRIPTION:
Reduction in beds coupled with the increased need for health care services has led to a supply and demand struggle or capacity management challenge for health care facilities. This is now recognized as a major public health issue. The impact is readily seen as overcrowding in emergency departments. At present 76% of hospitals' emergency departments (ETDs) are at or over capacity with 33% reporting ambulance diversions, the most common sign of overcapacity within a health care facility. Compounding the physical capacity problem is the "human capacity strain" as admitted patients remain in the ETD for prolonged periods waiting for beds. Delayed admission to patient care units significantly strains the financial resources, impedes "patient flow" ultimately impacting the quality of care, patient satisfaction and the "bottom line." Discharge before 11 am optimizes the availability of hospital beds to meet admission demands thereby avoiding a surge over capacity or "patient back log", ambulance diversions in ETD; the post anesthesia recovery unit, admissions office and critical care units. Conversely competing needs for the attending physician's physical presence off of the hospital premises; off of the unit (private practice and meetings) often delays patient discharge from before 11 am to the afternoon and evening.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Primary care physicians in internal medicine
* Primary care physicians/practice group with established discharge pattern after 11 am
* Primary care physicians/practice group with fast access digital subscriber line (DSL) 300 kilobytes per second
* Primary care physicians/practice group who have Hackensack Medical Center (HUMC) intranet access from pre-determined location

Exclusion Criteria:

* Non-English speaking patients
* Patients requiring acute level of care on the day of discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Timely patient discharge before 11 am
Patient satisfaction
Employee satisfaction

SECONDARY OUTCOMES:
Employee satisfaction
Physician satisfaction
Financial impact on medical center

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Feldman, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States